CLINICAL TRIAL: NCT01648985
Title: Diabetes in Minor Stroke and TIA, Glucose Tolerance and Haemostasis, a Long-term-follow-up Study and Intervention With Yoga
Brief Title: Diabetes in Minor Stroke/TIA, Glucose Tolerance and Haemostasis, a Long-term-follow-up Study and Intervention With Yoga
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Ann Charlotte Laska, Principal Investigator, Karolinska Institutet
Other Study IDs: catwil00
Record Dates: First submitted 2012-07-18; First posted 2012-07-25 (Estimated); Last update posted 2018-09-04 (Actual); Status verified 2018-08

CONDITIONS: Stroke; TIA
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Acute stroke and TIA patients: Cohort of acute stroke patients, admitted to the Stroke Unit Danderyd hospital 2010 - 2012
  Interventions: Other: Diabetes in stroke/TIA

INTERVENTIONS:
Other: Diabetes in stroke/TIA — Mostly no intervention. A small Group of the patients recieved Yoga

SUMMARY:
In acute stroke patients about 20 % have known diabetes. There is a doubled risk of recurrent stroke in diabetic patients. It has been shown that antiplatelet drugs are not as effective in diabetic patients as in non-diabetic patients. In acute stroke patients around 80 % have impaired glucose tolerance, which will improve after one month till about 60 %.

This study includes acute patients with minor stroke or TIA. They are followed up at one and six months and then at every six months for at least four years. The investigators perform an OGTT and haemostatic tests within the first days after onset and then at one month. Blood pressure, metabolic parameters, bodyweight, physical activity and diet are collected at each visit. The investigators give the patients information about lifestyle changes as needed.

As part of the study there is an interventional study, Medicine Yoga, an open randomized controlled study. Patients are randomized to 16 sessions of Yoga under professional instructions and a CD for home training or controls.

The aims of this study are to investigate glucose tolerance in acute stroke and TIA patients, and its relation to the different haemostatic variables. The importance of glucose tolerance, haemostatic variables and other risk factors (blood pressure, lipids, BMI,) on cardiovascular events will be investigated and the possibility to affect these risk factors by lifestyle changes and Yoga. The effect of different antiplatelet drugs will be investigated in relation to glucose tolerance.

DETAILED DESCRIPTION:
144 patients with minor stroke and TIA has been included in the study between 2010 and 2012. They have been follow for four years.

Two papers have been published on the results of the study. Lundström A, von Arbin M, Laska A C, Jörneskog G, Wallen NH. Glucose intolerance and insulin resistance as predictors of low platelet response to clopidogrel in patients with minor ischemic stroke or TIA. Platelets. 2013 Mar 25.341-49.

Lundström A, Wallén H, von Arbin M, Jörneskog G, Gigante B, Höeg Embrower K, Laurencikas E, Laska AC. Clopidogrel Resistance after Minor Ischemic Stroke or Transient Ischemic Attack is Associated with Radiological Cerebral Small-Vessel Disease. J Stroke Cerebrovasc Dis. 2015 Aug 21. pii: S1052-3057(15)00349-3

ELIGIBILITY:
Inclusion Criteria:

* Acute minor stroke and TIA patients able to perform OGTT within the first days after onset or having known diabetes.

Exclusion Criteria:

* Terminal disease

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute stroke and TIA patients screened from the stroke unit at Danderyd Hospital, Stockholm, Sweden
Sampling Method: Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Number of Stroke (fatal, non-fatal) | 4 years
  Stroke is defined on clinical ground with support by CT or MR scan

SECONDARY OUTCOMES:
Number of patients with Diabetes | 4years
  Diabetes is defined by HbA1c, OGTT,and fP-glucose

OTHER OUTCOMES:
Number of patients with Small Vessel Disease SVD | 4 years
  Diagnosed through CT-scan, Fazeca scale

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Daderyd Hospital, Stockholm, Sweden